CLINICAL TRIAL: NCT06382662
Title: Assessment of the Effect of Metaxalone 640 mg (M640) on Truck Driving Ability and Cognition Compared to Tizanidine 8 mg: A Prospective, Single-blind, Within-subject Pilot Study
Brief Title: Assess the Effect of Metaxalone 640 mg (M640) Compared to Tizanidine 8 mg on Truck Driving Ability and Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Sun Valley Arthritis Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PMDAC-01
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment
Keywords: Impaired driving
MeSH Terms: conditions — Cognitive Dysfunction | interventions — tizanidine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, single-blind, pilot study to assess degree of drowsiness, cognition, and driving risk following a single dose of oral metaxalone 640 mg (M640) compared to tizanidine 8 mg in healthy subjects.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- metaxalone m640 mg (Active Comparator): metaxalone micronized 640 mg tablet, single dose at Visit 2 or Visit 3
  Interventions: Drug: metaxalone m640
- tizanidine 8 mg (Active Comparator): tizanidine 8 mg tablet, single dose at Visit 2 or Visit 3
  Interventions: Drug: tizanidine

INTERVENTIONS:
Drug: metaxalone m640 — A single dose of micronize metaxalone 640 mg
  Other Names: Metaxalone 640
  Arms: metaxalone m640 mg
Drug: tizanidine — A single dose of tizanidine 8 mg
  Other Names: Zanaflex
  Arms: tizanidine 8 mg

SUMMARY:
Every participant will receive active study drug and one (1 )comparator, in two (2) stages, one after the other. Each drug will be taken one (1) time after a high fat meal. Vital signs and discussion of medications, illness or injury are considered safety assessments and will be discussed at every visit. There will be ( four (4) visits.

DETAILED DESCRIPTION:
Every participant will receive active study drug and one (1) comparator in two (2) stages, one after the other. Each drug will be taken one (1) time after a high fat meal. Vital signs and discussion of medications, illness or injury are considered safety assessments and will be discussed at every visit.

The Screening Visit will be followed by the Baseline (Visit 1) 1-14 days later. At the Baseline Visit participants will be given written tests to measure thinking process. You will also be asked to take a computer driving simulation test.

Visits 2 and 3 approximately one (1) week apart will be the dosing days after eating a high fat meal within 30 minutes. The testing from the Baseline Visit will be repeated at four (4) hours and 1.5 hours after dosing with comparator drug.

The End of Study safety visit will take place two (2) weeks later. Participants will be given discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* equal to or greater than 20 years old
* weight at least 120 pounds
* medically healthy
* able to eat a high fat meal

Exclusion Criteria:

* medications known to affect sleep-wake cycle
* current use of cimetidine
* current use of certain anti-depressants
* current us of certain antibiotics
* positive urine drug test for mind altering medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline, Standard Deviation of Lateral Position | Baseline, Visit 2 dosing, (day 1), Visit 3 dosing, (day 8)
  Using the One Motion GT Elite Mini- Simulator (SimGear) with Carnet Soft Driving Simulation Software
Change from baseline of participants' reasoning ability to recognize differences in six (6) computer generated shapes for 30 minutes | Visit 2 (Day 0), Visit 3 (Day 1). Visit 4 (Day 8)
  Creyos Cognitive Test

SECONDARY OUTCOMES:
Change from baseline of participants' subjective report of drowsiness on a 10-point scale | Visit 2 (Day 0), Visit 3 (Day 1). Visit 4 (Day 8)
  Karolinska Sleepiness Scale where 1 = extremely alert and 10 = extremely sleepy, can't keep awake
Percentage of participants unable to maintain Tandem Stand Position for more than 10 seconds (position 3 of the 4-Stage Balance Test) | Visit 2 (Day 0), Visit 3 (Day 1). Visit 4 (Day 8)
  Validated 4-Stage Balance Test after completion of an FDA standardized high-fat meal. Place one foot in front of the other, heel touching toes.
The number of product related adverse events experienced by participants from Visit 1 through Visit 4 | Baseline, Visit 2 (Day 0), Visit 3 (Day 1), Visit 4 (Day 8), Visit 4 (Day 15)
  Adverse and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: J C Lukban, DO, Study Director — Sponsor GmbH
Locations (1):
- Sun Valley Arthritis Center, Peoria, Arizona, United States